CLINICAL TRIAL: NCT02391675
Title: The Hasselt APPendicitis Immunology and Environmental Cohort STudy
Acronym: HAPPIEST
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hasselt University (Other)
Collaborators: Radboud University Medical Center (Other); Jessa Hospital (Other)
Responsible Party: Principal Investigator, prof. dr. Inge Gyssens, Prof. Dr., Hasselt University
Other Study IDs: 12.17/infect12.03
Record Dates: First submitted 2015-02-26; First posted 2015-03-18 (Estimated); Last update posted 2018-05-22 (Actual); Status verified 2018-05

CONDITIONS: Appendicitis
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Years
Biospecimen Retention: Samples With DNA — Whole blood, plasma, serum, appendix tissue, stool
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Appendicitis patients: Patients presenting with acute appendicitis

SUMMARY:
The Hasselt Appendicitis Immunology and Environmental Study (HAPPIEST) aims at characterizing factors that influence the development and severity of acute appendicitis. In a cohort of 300 patients and 300 controls, environmental factors as well as genetic make-up of the innate immune system, focusing mainly on pattern recognition, will be analyzed in order to gain insight in their relative importance in the pathology of appendicitis. Furthermore, populations of micro-organisms present in the gut of patients will be characterized, and the interaction between relevant micro-organisms and the innate immune system will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Acute appendicitis
* Appendectomy within 7 days after onset of symptoms
* Signed informed consent

Exclusion Criteria:

* Appendectomy 7 days or more after onset of symptoms
* Participation in any clinical investigational drug study within 4 weeks of screening
* Severe, life-threatening disease with a life expectancy of less than 2 months.

Ages: 5 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients are asked to participate after presenting with acute appendicitis at the emergency room of Jessa Ziekenhuis, Hasselt. If the patient fits the criteria, and informed consent is signed, the patient is included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 308 (Actual)
Dates: Start 2012-06; Primary Completion 2018-10 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Genetic susceptibility | Within 2 years after inclusion of the last patient
  DNA sample collected at inclusion

SECONDARY OUTCOMES:
Immunology composite outcome | within 4 years
  ex vivo peripheral blood mononuclear cell (PBMC) stimulation experiments
Environmental factors | Within 6 months after inclusion of the last patient
  Questionnaire filled in at inclusion

OTHER OUTCOMES:
Quality of life | 4-6 weeks after inclusion for appendicitis
  Questionnaire at outpatient visit

CONTACTS AND LOCATIONS:
Overall Officials: Inge C Gyssens, MD PhD, Principal Investigator — Hasselt University
Locations (2):
- Jessa Ziekenhuis, Hasselt, Limburg, Belgium
- Radboud University Medical Center, Nijmegen, Gelderland, Netherlands

REFERENCES:
- [Background] Stappers MH, Thys Y, Oosting M, Plantinga TS, Ioana M, Reimnitz P, Mouton JW, Netea MG, Joosten LA, Gyssens IC. Polymorphisms in cytokine genes IL6, TNF, IL10, IL17A and IFNG influence susceptibility to complicated skin and skin structure infections. Eur J Clin Microbiol Infect Dis. 2014 Dec;33(12):2267-74. doi: 10.1007/s10096-014-2201-0. Epub 2014 Jul 15. PMID 25022448
- [Background] Stappers MH, Thys Y, Oosting M, Plantinga TS, Ioana M, Reimnitz P, Mouton JW, Netea MG, Joosten LA, Gyssens IC. TLR1, TLR2, and TLR6 gene polymorphisms are associated with increased susceptibility to complicated skin and skin structure infections. J Infect Dis. 2014 Jul 15;210(2):311-8. doi: 10.1093/infdis/jiu080. Epub 2014 Feb 6. PMID 24511099
- [Background] Rivera-Chavez FA, Peters-Hybki DL, Barber RC, Lindberg GM, Jialal I, Munford RS, O'Keefe GE. Innate immunity genes influence the severity of acute appendicitis. Ann Surg. 2004 Aug;240(2):269-77. doi: 10.1097/01.sla.0000133184.10676.26. PMID 15273551
- [Background] Schnitzler F, Friedrich M, Wolf C, Angelberger M, Diegelmann J, Olszak T, Beigel F, Tillack C, Stallhofer J, Goke B, Glas J, Lohse P, Brand S. The NOD2 p.Leu1007fsX1008 mutation (rs2066847) is a stronger predictor of the clinical course of Crohn's disease than the FOXO3A intron variant rs12212067. PLoS One. 2014 Nov 3;9(11):e108503. doi: 10.1371/journal.pone.0108503. eCollection 2014. PMID 25365249
- [Derived] Peeters T, Penders J, Smeekens SP, Galazzo G, Houben B, Netea MG, Savelkoul PH, Gyssens IC. The fecal and mucosal microbiome in acute appendicitis patients: an observational study. Future Microbiol. 2019 Jan;14:111-127. doi: 10.2217/fmb-2018-0203. Epub 2019 Jan 21. PMID 30663346